CLINICAL TRIAL: NCT00212433
Title: Multidetector-row CT Colonography: Optimisation of Reduced Bowel Preparation Regimes and Diagnostic Performance in Comparison to Colonoscopy
Brief Title: Optimisation and Performance of Reduced Preparation CT Colography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: St Mark's Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 04/Q0405/CT2
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Patients With Potential Colorectal Neoplasia
Keywords: colorectal neoplasia; CT colonography; faecal tagging
MeSH Terms: interventions — Barium Sulfate

INTERVENTIONS:
Drug: Tagitol V, Lo So, Readi-Cat 2

SUMMARY:
To ascertain which of four combinations of low residue diet, reduced laxative dose and oral contrast agent is best tolerated by patients and optimally prepares the colon prior ro CT colonography

DETAILED DESCRIPTION:
CT colonography has been shown to be accurate in detection of colorectal neoplasia in enriched patient populations and is generally preferred by patients to conventional endoscopy and barium enema. It is advocated as an acceptable alternative for colorectal cancer screening and is increasingly used in the investigation of symptomatic patients. Ideally, like conventional colonoscopy, CT colonography requires a clean colon, free of residual stool and fluid. There is however good evidence that the arduous bowel purgation regimes required may produce adverse effects such as electrolyte imbalance, and are more detrimental to overall patient experience and compliance than any subsequent investigation. An ability to perform CT colonography with reduced bowel purgation, whilst maintaining acceptable diagnostic accuracy, would undoubtedly make the technique a more attractive proposition both for population screening and investigation of symptomatic patients.

Interest has been generated in the use of orally ingested dilute barium or ionated contrast medium prior ro CT colonography to "label" or "tag" residual fluid or faecal matter reduced laxative. Such oral contrast agents are highly attenuating to X-rays such that labeled residual bowel contents appear white on CT scanning and are readily distinguished from true colonic pathology.

Despite the early promise of a few limited studies, there is no consensus as to the optimum oral contrast type, dose and concentration. Anecdotally barium tends to best label solid residue whereas iodinated contrast best labels fluid, but this assumption has not been proven. Furthermore it is known that iodinated contrast tends to draw fluid into the bowel, producing a wet colon, which may not be suited to CT colonography. However, this indrawing of fluid by iodinated contrast such as gastrograffin produces a mild laxative effect, which may obviate the need for further formal purgation.

The study aims to establish the optimum reduced preparation-tagging regimen, establish patient experience and document diagnostic performance compared to conventional colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are under investigation for suspected colonic neoplasia and over 50 years old:

  1. Symptomatic patients eg. change in bowel habit, rectal bleeding etc.
  2. Polyp surveillance
  3. Strong family history
  4. suspected neoplasia on previous investigation (e.g. barium enema)

Exclusion Criteria:

* patients under 50 patients undergoing surveillance for inflammatory bowel disease (due to poor diagnostic use of CT colonography in this specific patient cohort)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-07; Study Completion 2006-02

PRIMARY OUTCOMES:
Which of four combinations of low residue diet, reduced laxative dose and oral contrast agent is best tolerated by patients and optimally prepares the colon prior ro CT colonography

SECONDARY OUTCOMES:
to compare the diagnostic performance of CT colonography after reduced bowel preparation and faecal tagging with conventional colonoscopy in patients undergoing both procedures

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Taylor, MD, Principal Investigator — St Mark's Hospital, North West London NHS Trust; & University College Hospital
Locations (3):
- United Kingdom (3):
  - St Mark's Hospital, North West London Hospitals NHS Trust, London, Middlesex
  - University College Hospital, London
  - Oxford Radcliffe Hospital NHS Trust, Oxford